CLINICAL TRIAL: NCT00551954
Title: Effects of Acarbose on Endothelial Function After a Mixed Meal in Newly Diagnosed Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIDA a4
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 20 weeks of treatment with acarbose (100 mg t.i.d.)
  Interventions: Drug: acarbose
- 2 (Placebo Comparator): 20 weeks of treatment with placebo (one tablet t.i.d.)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: acarbose — 100 mg (tablets) t.i.d.
  Arms: 1
Drug: placebo — one tablet t.i.d.
  Arms: 2

SUMMARY:
Endothelial dysfunction (ED) has been suggested as a possible causal link between postprandial hyperglycemia and cardiovascular events in patients with type 2 diabetes. Recent trials demonstrated a reduction of cardiovascular events by treatment with the alpha glucosidase inhibitor acarbose - a drug which mainly reduces postprandial glucose excursions. We were interested whether patients with newly diagnosed type 2 diabetes showed postprandial ED and if so whether acarbose was able to improve this condition.

ELIGIBILITY:
Inclusion Criteria:

* age 35-75 years
* type 2 diabetes (newly diagnosed)
* well glycemic control (HbA1c </= 8.1)
* leucocyte count > 6.2 or hs CrP > 1

Exclusion Criteria:

* hs CrP > 10
* type 1 diabetes
* previous treatment with antidiabetic drugs

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-07; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
forearm blood flow assessed by forearm occlusion plethysmography after a mixed meal | at baseline and after 20 weeks of treatment

SECONDARY OUTCOMES:
forearm blood flow assessed by forearm occlusion plethysmography in the fasting state, plasma glucose excursion in response to the mixed meal, insulin levels in response to the mixed meal, triglyceride levels in response to the mixed meal | at baseline and after 20 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Markolf Hanefeld, PhD, Principal Investigator — Center for Clinical Studies, Fiedlerstr. 34, 01307 Dresden, Germany